CLINICAL TRIAL: NCT04110899
Title: Paratracheal Force Required for Occluding the Upper Esophagus in Anesthetized and Paralyzed Patients
Brief Title: Paratracheal Force Required for Occluding the Upper Esophagus
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: SMG-SNU Boramae Medical Center (Other)
Responsible Party: Principal Investigator, Jin-Young Hwang, Associate professor, SMG-SNU Boramae Medical Center
Model: Sequential | Masking: None | Purpose: Prevention
Other Study IDs: 2019-6209
Record Dates: First submitted 2019-09-26; First posted 2019-10-01 (Actual); Last update posted 2020-06-19 (Actual); Status verified 2020-06

CONDITIONS: Anesthesia Intubation Complication

STUDY DESIGN:
Intervention Model Description: Paratracheal force for occluding the upper esophagus is evaluated using the up-and-down sequential method.
Masking Description: Participant: masked because the intervention is applied after anesthesia induction Care provider who inserts an esophageal stethoscope under a certain paratracheal force: masked. The amount of applied paratracheal force is not shown to this investigator
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Different paratracheal force (Experimental): Esophageal occlusion is assessed by inserting an esophageal stethoscope under different paratracheal forces.
  Interventions: Other: Application of paratracheal force

INTERVENTIONS:
Other: Application of paratracheal force — An esophageal stethoscope is inserted into the upper esophagus under the application of different paratracheal force in anesthetized and paralyzed patients.

SUMMARY:
In this study, the median paratracheal force for occluding the upper esophagus are evaluated in anesthetized and paralyzed patients using the up-and-down technique.

ELIGIBILITY:
Inclusion Criteria:

* patients who are scheduled for elective surgery under general anesthesia

Exclusion Criteria:

* diseases or anatomical abnormalities in the neck, larynx, pharynx or esophagus
* aspiration tendency
* history of carotid artery diseases or cerebrovascular diseases
* suspicious of thrombus in carotid artery on ultrasonographic examination

Min Age: 20 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 47 (Actual)
Dates: Start 2020-03-03 (Actual); Primary Completion 2020-06-10 (Actual); Study Completion 2020-06-10 (Actual)

PRIMARY OUTCOMES:
Median paratracheal force | During 1 min after the completion of anesthesia induction
  Esophageal occlusion is evaluated under different paratracheal force by inserting the esophageal stethoscope

SECONDARY OUTCOMES:
The 95% paratracheal force | During 1 min after the completion of anesthesia induction
  Esophageal occlusion is evaluated under different paratracheal force by inserting the esophageal stethoscope

CONTACTS AND LOCATIONS:
Locations (1):
- SMG-SNU Boramae Medical Center, Seoul, South Korea